CLINICAL TRIAL: NCT02561910
Title: Effectivity of Laparoscopic Inguinal Hernia Repair (TAPP) in Daily Clinical Practice - Early and Long-term Results
Status: Completed | Type: Observational
Sponsor: Hernia Center Rottenburg (Other)
Responsible Party: Principal Investigator, Prof.Dr. Reinhard Bittner, Director, Hernia Center Rottenburg
Other Study IDs: HerniaCR
Record Dates: First submitted 2015-09-25; First posted 2015-09-28 (Estimated); Last update posted 2015-09-28 (Estimated); Status verified 2015-09

CONDITIONS: Unilateral Inguinal Hernia With Gangrene and Obstruction
Keywords: Inguinal hernia repair; laparoscopic inguinal hernia repair; TAPP
MeSH Terms: conditions — Bites and Stings

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Laparoscopic hernia repair — Preperitoneal mesh implantation because of inguinal hernia disease using the laparoscopic technique

SUMMARY:
The effectiveness of laparoscopic inguinal hernia repair still remains unclear. During a one year period a total of 1208 inguinal hernias in 952 patients were consecutively operated using the laparoscopic technique by a total of 11 general surgeons in daily clinical routine.

Laparoscopic hernia repair in the TAPP technique seems to have the potential to become the standard procedure in inguinal hernia repair in future.

DETAILED DESCRIPTION:
Objective:

Hernia repair is the most frequent operation in general surgery worldwide, but about 25 years after the advent of minimal invasive surgical techniques the effectiveness of laparoscopic inguinal hernia repair still remains unclear.

Methods:

All patients admitted to the hospital for surgery of an inguinal hernia during a one year period were prospectively documented and included in a follow-up study. The follow-up was performed at least 5 years after surgery and consisted of a clinical examination, ultrasound investigation and a questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* All patients fit for general anesthesia and presenting an inguinal hernia.

Exclusion Criteria:

* Not fit for general anesthesia, young age (>21 years), not wanting a mesh.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients admitted for hernia surgery during a one year period (n=928) were operated exclusively in TAPP technique and were assigned to follow-up.
Sampling Method: Non-Probability Sample
Enrollment: 952 (Actual)
Dates: Start 2000-01; Primary Completion 2008-12 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
The primary outcome of the trial was recurrence of a hernia within five years after the repair. | 5 years

SECONDARY OUTCOMES:
The secondary outcome was chronic pain. | 5 years
  Chronic pain was measured by VAS scale

CONTACTS AND LOCATIONS:
Overall Officials: Reinhard Bittner, M.D., Principal Investigator — Hernia Center Rottenburg
Locations (1):
- Hernia Center, Rottenburg, Germany

REFERENCES:
- [Background] Cavazzola LT, Rosen MJ. Laparoscopic versus open inguinal hernia repair. Surg Clin North Am. 2013 Oct;93(5):1269-79. doi: 10.1016/j.suc.2013.06.013. PMID 24035088